CLINICAL TRIAL: NCT02827461
Title: Heritability of Sleep Homeostasis in Twins
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Allan Pack, Co-Project Leader, University of Pennsylvania
Other Study IDs: 704868; P50HL060287 (NIH); P01HL094307 (NIH)
Record Dates: First submitted 2016-06-27; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Hereditability of Sleep Homeostasis in Twins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and DNA samples will be identified by a bar-coding system. This will only be able to be matched to the subject ID using a secure computer database to which only the Principal Investigator will have access.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MZ: Monozygotic twins
- DZ: Dizygotic twins

SUMMARY:
The purpose of this study is to understand the hereditability of sleep homeostasis, i.e., drive for sleep by looking at monozygotic and dizygotic twins.

DETAILED DESCRIPTION:
Excessive daytime sleepiness is a prevalent problem in our society associated with an increased risk of vehicular crashes and industrial accidents. Sleepiness is, in part, determined by fundamental biology relating to sleep homeostasis, i.e., the rate of accumulation of the pressure for sleep during wakefulness. A differential susceptibility to sleep deprivation is reported in normal subjects with large intraindividual differences in the degree of functional impairment produced by the same duration of sleep. Genetics are likely to play an important role in sleep homeostasis as shown by recent studies in inbred mouse strains, but whether genetics plays any role in humans and, if so, the magnitude of this role, is unknown. This proposal is based on the hypothesis that sleep homeostasis is a heritable trait in humans. Given the complexity of phenotyping to study sleep homeostasis, the investigators propose that studying differences in the variances of the phenotype between monozygotic and dizygotic twins is the optimal approach to estimate heritability of sleep homeostasis. The investigators will assess sleep homeostasis in 80 pairs of monozygotic and 80 pairs of dizygotic twins by quantifying the increase in delta power during recovery sleep following sleep deprivation and the increase in theta power during the period of prolonged wakefulness. Subjects will be recruited using the PennTwins Cohort, a population-based cohort of about 1,800 twin pairs. If heritability of sleep homeostasis is shown, this EEG-based phenotyping strategy could not be easily applied to the larger scale population studies that will be required to assess underlying genetic variants. Thus, part of the overall strategy is to evaluate, and potentially validate, other approaches to phenotyping that are less physiologically rigorous but are more easily applied to a larger number of subjects. Therefore, as a subsidiary goal, the investigators will also estimate heritability of performance lapses during prolonged wakefulness as a surrogate method to assess sleep homeostasis. The investigators will particularly determine whether the differences in the measures based on our physiological intensive phenotypes between pairs of dizygotic twins are reflected in differences in this phenotyping approach that is simpler to perform. Such a result would indicate that this simpler method could be used in larger scale population studies, and will be part of future strategies to elucidate genetic variants determining sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Being a twin with a twin of same gender
* Age between18 and 55 years

Exclusion Criteria:

All exclusion criteria apply to both members if one twin has any exclusion. The exclusion criteria include the following:

* Previous diagnosis of sleep disorder, e.g., narcolepsy, obstructive sleep apnea; presence of conditions that could interrupt sleep, e.g., chronic pain, asthma, arthritis; presence of fibromyalgia; previous clinical diagnosis of major depression; history of alcoholism or drug abuse; any medical disorder that limits their ability to participate in protocol;
* Use of sedative/hypnotics to promote sleep; use of stimulants, e.g., methylphenidate; use of modafinil; excessive use of caffeine (>500 mg/day); use of psychoactive medications, e.g., antidepressants;
* Shift-work; regular travel across time zones, in particular in the 6 weeks prior to study enrollment; irregular sleep/wake patterns. (This will be assessed prior to in-depth phenotyping by measurement of rest/activity at home (see further below);
* Inability to comprehend English (questionnaires and consent form are in English),
* The study will exclude women who are pregnant or perimenopausal but include women who are postmenopausal without hot flashes, or premenopausal.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be healthy MZ and DZ twins of the same gender between 18 years and 55 years of age.
  The investigators will not exclude any specific racial or ethnic group. African-American twins currently represent 3.8% of the PennTwins Cohort, i.e., 68 twin pairs. The investigators plan to oversample this group. The study design calls for 8 MZ and 8 DZ African-American twins to match the demographics of the population. There are currently no data that the phenotype being studied is affected by race or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Measure heritability of sleep by increase in electroencephalographic slow-wave activity | Through study completion, 4-6 weeks
  The investigators will measure this during recovery NREM sleep following a period of prolonged wakefulness and the increase in theta power during the prolonged wakefulness period

REFERENCES:
- [Derived] Gao X, Azarbarzin A, Keenan BT, Ostrowski M, Pack FM, Staley B, Maislin G, Pack AI, Younes M, Kuna ST. Heritability of Heart Rate Response to Arousals in Twins. Sleep. 2017 Jun 1;40(6):zsx055. doi: 10.1093/sleep/zsx055. PMID 28431171